CLINICAL TRIAL: NCT01553656
Title: Phase 1 Multiple Ascending Dose Study of XL184 Monotherapy in Japanese Subjects With Advanced or Metastatic Solid Tumors
Brief Title: Dose-Finding Study of Cabozantinib (XL184) in Japanese Subjects With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XL184-014
Record Dates: First submitted 2012-03-09; First posted 2012-03-14 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Solid Tumors; Cancer; NSCLC
Keywords: Advanced cancer; Metastatic; NSCLC
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — cabozantinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cabozantinib capsules and tablets (Experimental): Subjects will be enrolled in cohorts at different dose levels in order to determine the maximum tolerated dose of cabozantinib. Initially, subjects enrolled will receive the capsule formulation; other subjects will receive the tablet formulation.
  Interventions: Drug: cabozantinib capsules; Drug: cabozantinib tablets

INTERVENTIONS:
Drug: cabozantinib capsules — cabozantinib capsules administered as 25-mg and 100-mg strengths once-daily until disease progression
  Other Names: XL184
Drug: cabozantinib tablets — cabozantinib tablets administered as 20-mg and 60-mg strengths once-daily until disease progression
  Other Names: XL184

SUMMARY:
The purpose of this study is to evaluate the safety profile, tolerability, pharmacokinetics (PK), pharmacodynamics, pharmacogenomic (PGX) and preliminary efficacy following daily oral doses of cabozantinib (XL184) in Japanese patients with advanced or metastatic solid tumors. Also, the effect of XL184 in the treatment of non-small cell lung cancer (NSCLC) patients with various activating mutations will be evaluated at the recommended Phase 2 dose.

ELIGIBILITY:
Select Inclusion Criteria:

* Subjects with advanced or metastatic solid tumors for whom the standard of care is ineffective or inappropriate.
* NSCLC expansion cohort subjects must have confirmed NSCLC (Stage IIIb or IV) and documented activating mutations.
* At least 4 weeks must have elapsed from the last anti-cancer therapy. At least 6 weeks for nitrosoureas, mitomycin C and liposomal doxorubicin.
* Have adequate bone marrow function, adequate liver function, and adequate renal function.
* Sexually active subjects (men and women of child-bearing potential (WOCBP)) must agree to use medically accepted barrier methods of contraception (eg, male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used. All subjects of reproductive potential must agree to use both a barrier method and a second method of birth control. Women of childbearing potential (WOCBP) must have a negative pregnancy test at screening.

Select Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastasis, or active CNS metastasis requiring medication.
* WOCBP who are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for the entire study period and for 4 months after the last dose of investigational product.
* Women who are pregnant or breastfeeding.
* Sexually active fertile men not using effective birth control for the entire study period and for 4 months after the last dose of investigational product if their partners are WOCBP.
* Subjects who have uncontrolled intercurrent illness including, but not limited to, infection requiring systemic therapy, symptomatic congestive heart failure, uncontrolled hypertension, uncontrolled angina pectoris, uncontrolled peptic ulcer, cardiac arrhythmia requiring medication.
* Subjects who are HIV antibody positive, HBs antigen positive, and/or HCV antibody positive.
* Subjects with body cavity fluid retention which requires drainage.
* Subjects with any major surgery within 8 weeks prior to study enrollment.
* Subjects with major unhealed wounds or fracture.
* Subjects with a history or concurrent diagnosis of gastrointestinal perforation.
* Subjects with evidence of bleeding tendency or coagulopathy.
* Subjects with a history of thromboembolism.
* Subjects with a history of or concurrent pancreatitis.
* Exposure to any investigational drug within 30 days of enrollment.
* Subjects receiving radiation therapy or treatment with radionuclides within 6 to 2 weeks before first dose of XL184.
* NSCLC expansion cohorts: subjects must not be diagnosed with another malignancy within 2 years before first dose of XL184.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose | Assessed in the clinic on Days 1 through 29
  To establish the MTD and recommended Phase 2 dose (or dose range as appropriate) of XL184 when administered orally on a once daily schedule in subjects with advanced or metastatic solid tumors.

SECONDARY OUTCOMES:
Safety and tolerability of XL184 | From study start to October 2014
  Safety and tolerability of multiple doses of XL184 administered orally on a daily basis. Assessed from informed consent until at least 30 days after discontinuation.
Plasma Pharmacokinetics | Assessed in the clinic from Day 1 through Day 29
  Assess plasma pharmacokinetics of daily oral administration of XL184 from Treatment Day 1 to Day 29.
Tumor response (preliminary anti-tumor activity) | Study start to October 2014
  Assess tumor response after repeated administration of XL184 from screening until discontinuation. Assessed as best overall response by cohort by radiological response defined by RECIST criteria.

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - The Cancer Institute Hospital of the Japanese Foundation for Cancer Research (JFCR), Ariake, Koto
  - National Cancer Center Hospital, Chuo-ku, Tokyo

REFERENCES:
- [Derived] Nokihara H, Nishio M, Yamamoto N, Fujiwara Y, Horinouchi H, Kanda S, Horiike A, Ohyanagi F, Yanagitani N, Nguyen L, Yaron Y, Borgman A, Tamura T. Phase 1 Study of Cabozantinib in Japanese Patients With Expansion Cohorts in Non-Small-Cell Lung Cancer. Clin Lung Cancer. 2019 May;20(3):e317-e328. doi: 10.1016/j.cllc.2018.12.018. Epub 2018 Dec 31. PMID 30718102